CLINICAL TRIAL: NCT01333670
Title: Efficacy of Prontosan Solution on Chronic Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Associazione Infermieristica per lo studio delle Lesioni Cutanee (Other)
Collaborators: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AISLeC-001
Record Dates: First submitted 2011-04-06; First posted 2011-04-12 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2011-04

CONDITIONS: Pressure Ulcer; Chronic Wound Care; Wound Cleansing
MeSH Terms: conditions — Pressure Ulcer | interventions — Isotonic Solutions; Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prontosan wound irrigation solution (Experimental)
  Interventions: Device: Prontosan wound irrigation solution
- Standard care (Active Comparator)
  Interventions: Drug: Isotonic solution (saline or lactated ringer)

INTERVENTIONS:
Device: Prontosan wound irrigation solution — * cleansing wound bed at change with Prontosan Wound Irrigation solution (syringe 20-30 ml, needle 19-20 G)
  * positioning of sterile gauze dressing impregnated with Prontosan Wound Irrigation solution on the wound for 10 minutes
  * dressing with Prontosan Wound Irrigation solution
  Arms: Prontosan wound irrigation solution
Drug: Isotonic solution (saline or lactated ringer) — * cleansing wound bed at change with isotonic solution (syringe 20-30 ml, needle 19-20 G)
  * positioning of sterile gauze dressing impregnated with isotonic solution on the wound for 10 minutes
  * dressing with isotonic solution
  Arms: Standard care

SUMMARY:
The purpose of this study is to evaluate the efficacy of Prontosan® Wound Irrigation Solution compared with standard isotonic solution on infammation reduction and wound bed cleansing of chronic pressure or vascular leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged at least 18 with Pressure ulcer stage 2-3 NPUAP (National Pressure Ulcer Advisory Panel 1989)or subcutaneous vascular ulcer with inflammation and/or biofilm and/or slough
* Braden index at baseline>=10
* Ulcer area<80 cm2
* Ability to give an informed consent

Exclusion Criteria:

* Braden index at baseline<10
* Current therapy with corticosteroids or immunosuppressor or radiotherapy
* Sensitivity to any of the components of Prontosan® Solution
* Diabetic foot ulcer
* Current use of local antiseptics on the wound bed
* Previous recruitment of another ulcer in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reduction of necrotic tissue (Pressure Sore Status Tool-PSST) | From basaline visit to the final visit, that is between a minimum of 1 visit (10 days later) or a maximum of 4 visits (1 month later, weekly)
Reduction of inflammatory tissue(Pressure Sore Status Tool-PSST) | From basaline visit to the final visit, that is between a minimum of 1 visit (10 days later) or a maximum of 4 visits (1 month later, weekly)

SECONDARY OUTCOMES:
Frequency of wound dressing (clinical score) | From basaline visit to the final visit, that is between a minimum of 1 visit (10 days later) or a maximum of 4 visits (1 month later, weekly)

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Azienda Ospedaliera Ospedale di Circolo di Busto Arsizio, Busto Arsizio, Milan
  - Home nursing assistance, Florence
  - Policlinico San Matteo, Pavia
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Trieste
  - Azienda Ospedaliero Universitaria San Giovanni Battista, Turin
  - Ospedale di Circolo-Fondazione Macchi, Varese